CLINICAL TRIAL: NCT04664998
Title: Alignment of PrEP Use With HIV Risk in Young Women and Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Makerere University (Other); MU-JHU CARE (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Renee Heffron, Official Title: Associate Professor, Global Health and Epidemiology Affiliation: University of Washington, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008057; R21HD098923 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2020-12-11 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Pre-Exposure Prophylaxis; Sexually Transmitted Diseases, Bacterial; HIV Infections
Keywords: HIV acquisition; HIV risk; PrEP adherence
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; HIV Infections

STUDY DESIGN:
Intervention Model Description: The two groups are male participants enrolled in the Align study, and their sexual partners enrolled in the parent study, Kampala Women's Bone study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male participants (Active Comparator): Male participants whose partners are enrolled in the parent study (Kampala Women's Bone study). All male participants will undergo the same study procedures at each visit, such as HIV and STI testing, and urine tenofovir testing if on PrEP.
  Interventions: Drug: Daily oral PrEP
- Female participants (Active Comparator): Female participants from the parent study (Kampala Women's Bone study) will be enrolled to recruit their male sexual partner(s). All female participants will receive HIV testing, STI testing, and urine tenofovir testing (if on PrEP) at quarterly visits.
  Interventions: Drug: Daily oral PrEP

INTERVENTIONS:
Drug: Daily oral PrEP — All participants will be offered daily oral PrEP at each visit
Drug: Daily oral PrEP — All participants will be offered daily oral PrEP at each visit.

SUMMARY:
Oral pre-exposure prophylaxis (PrEP) is a recommended component of combination HIV prevention and its availability is rising through demonstration projects and full-scale national programs. In sub-Saharan Africa, young women are a priority population for HIV prevention and targeted to initiate PrEP, given their high HIV incidence rates and promising success from a strategy that can be used without the engagement of male partners. A key question in the field is whether young women using PrEP have ongoing HIV risk and adhere to PrEP sufficiently to have protection from HIV when they have condomless sex with HIV-infected partners. The only true way to know whether a heterosexual woman is sexually exposed to HIV or has a partner with high HIV risk is to test for HIV and STIs in her male partner(s) and quantify HIV viral levels, if any are detected. Yet engaging men in clinic-based HIV testing is challenging. More recent efforts have focused on using HIV self-testing kits to respond to demands on men's time and reluctance to seeking preventive healthcare. The availability of PrEP also provides a new incentive for men to test.

By leveraging an ongoing study of bone health with concurrent use of PrEP and injectable DMPA (often known as Depo Provera® or depot medroxyprogesterone acetate), we have opportunity to engage a new cohort of young men and objectively measure HIV and common STIs in these young men and link the results to women's use of PrEP. The primary objective of this study is to determine whether young women's adherence to PrEP aligns with the HIV status and risk of their male partners. To address its primary objectives, this study will leverage: 1) an ongoing study among young women and 2) a novel cohort of young men who are current sexual partners of the young women in the ongoing study to objectively measure PrEP use, HIV, and HIV factors related to HIV risk. This study will provide a framework for understanding how and when young women and men decide to take PrEP, estimate the proportion of women that are benefitting from HIV protection when they have male partners with or at high risk of acquiring HIV, and provide a novel opportunity to engage young men in PrEP delivery and as supporters of women's PrEP use.

DETAILED DESCRIPTION:
The proposed research will engage a new cohort of young men, whose female partners are already engaged in the Kampala Women's Bone Study. Women in the Kampala Women's Bone Study will be invited to engage in this novel study to recruit their male partners. Women's HIV risk is directly related to the HIV status and risk of their male sexual partners and thus, we will leverage our ongoing cohort of KWBS young women to recruit their male sexual partners for a new men's study. Men will be offered PrEP, diagnostic STI testing and treatment, and followed for 6 months to assess PrEP continuation and STIs. Men's data will be linked to data from their female sex partners in the parallel KWBS study to determine whether women's PrEP use aligns with HIV risk and exposure.

B. Study Aims Aim 1. To determine whether young women's adherence to PrEP aligns with the HIV status of their male partners Men engaging in this study will have HIV testing at enrollment, month 1 and quarterly for up to 6 months. Results from this testing will be linked to data from the participant's female sex partner that characterize her PrEP use to determine whether her PrEP use aligns with his HIV status.

Aim 2. To determine whether young women's adherence to PrEP aligns with the HIV risk of their male partners Men engaging in this study will have testing for common curable STIs (Chlamydia trachomatis and Neisseria gonorrhoeae) at enrollment, month 1 and quarterly for up to 6 months. Results from this testing will be linked to data from the participant's female sex partner that characterize her PrEP use to determine whether her PrEP use aligns with his HIV risk (defined by the results from his STI testing).

Aim 3. To determine whether young men's adherence to PrEP aligns with the HIV status and risk of their female partners We will offer PrEP to HIV-negative men enrolled in this study and track PrEP initiation, refills, and adherence to PrEP (based on self-report and drug levels). The frequency of high PrEP adherence will be compared among men with female partners infected and uninfected with HIV or another STI.

C. Primary exposure The primary exposure is male infection with HIV (Aim 1), NG or CT (Aim 2) and female infection with HIV, NG, or CT (Aim 3).

D. Primary outcomes The primary outcome will be PrEP used by women with sufficient daily adherence to confer HIV protection (6-7 doses in the past week or TFV ≥40ng/mL) for periods when women are dispensed PrEP. When PrEP is not dispensed, the TFV level will be assigned as 0 ng/mL.

For Aim 3, the primary outcome will be PrEP used by men with sufficient daily adherence to confer HIV protection (4 doses in the past

ELIGIBILITY:
Inclusion Criteria:

* Men ages ≥18
* Has a female sexual partner enrolled in the Kampala Women's Bone Study
* Willing and able to provide informed consent

Exclusion Criteria:

* Has any other condition that would preclude the ability to provide informed consent, make study participation unsafe, complicate the interpretation of study findings or otherwise interfere with achievement of the study objectives, in the investigator's discretion.

Eligibility for women:

Inclusion criteria:

* Participating in the Kampala Women's Bone Study
* Willing to talk with male sex partners about the new study for men and refer men for study recruitment

Exclusion criteria:

* Has concerns about potential social harm stemming from anticipated conversations with male sex partners about the new study for men such that study staff would discourage the women from participation
* Investigator discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Heffron, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu L, Ssebuliba T, Muwonge TR, Bambia F, Stein G, Nampewo O, Sapiri O, Goetz BJ, Penrose KJ, Parikh UM, Mujugira A, Heffron R. Alignment of PrEP Use With Potential HIV Exposure in Young Women and Men in Uganda. J Acquir Immune Defic Syndr. 2025 Apr 1;98(4):326-333. doi: 10.1097/QAI.0000000000003573. Epub 2025 Feb 19. PMID 39630076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Male Participants | Female Participants
Started | 124 | 88
Completed | 124 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Male Participants | Female Participants | Total
Number analyzed (Participants) | 124 | 88 | 212
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23.5 [21 to 26] | 20.6 [19.5 to 22] | 22 [20.2 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 88 | 88
  Male | 124 | 0 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 124 | 88 | 212
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 124 | 88 | 212
PrEP dispensation at first visit [Count of Participants; unit: Participants] | 75 | 83 | 158

OUTCOME MEASURES:

1. Primary Outcome: Visits With PrEP Dispensation to Female Study Participants Reporting Sexual Behaviors or STI Symptoms
Description: Percentage of visits when PrEP was dispensed to female study participants at a visit when they self-reported sexual behaviors indicating potential HIV exposure (condomless sex, multiple sexual partners, Y-chromosome detection) or STI symptoms
Time Frame: Six months of study participation
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Groups:
- % Female Participant Visits When PrEP Dispensed: Female participants from the parent study (Kampala Women's Bone study) will be enrolled to recruit their male sexual partner(s). All female participants will receive HIV testing, STI testing, and urine tenofovir testing (if on PrEP) at quarterly visits.
  Daily oral PrEP: All participants will be offered daily oral PrEP at each visit
  Daily oral PrEP: All participants will be offered daily oral PrEP at each visit.
Arm/Group | % Female Participant Visits When PrEP Dispensed
Number analyzed (Participants) | 88
Number analyzed (Visits) | 332
Visits | 211

2. Primary Outcome: Visits With PrEP Dispensation to Male Study Participants Reporting Sexual Behaviors or STI Symptoms
Description: Percentage of visits when PrEP was dispensed to male study participants at a visit when they self-reported sexual behaviors indicating potential HIV exposure (condomless sex, multiple sexual partners) or STI symptoms
Time Frame: Six months
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Groups:
- % Male Participant Visits When PrEP Dispensed: Male participants whose partners are enrolled in the parent study (Kampala Women's Bone study). All male participants will undergo the same study procedures at each visit, such as HIV and STI testing, and urine tenofovir testing if on PrEP.
  Daily oral PrEP: All participants will be offered daily oral PrEP at each visit
  Daily oral PrEP: All participants will be offered daily oral PrEP at each visit.
Arm/Group | % Male Participant Visits When PrEP Dispensed
Number analyzed (Participants) | 124
Number analyzed (Visits) | 241
Visits | 151

ADVERSE EVENTS:
Time Frame: Six months
Description: Adverse event data were reported spontaneously by participants and not routinely collected.
Arm/Group | Male Participants | Female Participants
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/88
Other Adverse Events (participants affected / at risk) | 0/124 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04664998/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04664998/ICF_001.pdf